CLINICAL TRIAL: NCT07343921
Title: Comparison of Lung Function in Post-CABG Patients Administered Supervised and Non-supervised Post-operative Incentive Spirometry: a Quasi-experimental Study
Brief Title: Supervised vs Non-Supervised Incentive Spirometry After CABG
Acronym: SIS-CABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Arnengsih Nazir, Principal Investigator, Universitas Padjadjaran
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IKFR-202502.01; DP.04.03/D.XIV.6.5/77/2024 (Other: Komite Etik Penelitian RSUP Dr. Hasan Sadikin Bandung)
Record Dates: First submitted 2025-12-19; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pulmonary Function Impairment
Keywords: CABG; incentive spirometry; pulmonary function; supervision; postoperative care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Incentive Spirometry (SIS) (Experimental): Participants perform incentive spirometry exercises twice daily for 3 days under direct supervision. The supervisor observes the technique, provides corrections, answers questions, and ensures adherence to the prescribed exercise regimen.
  Interventions: Procedure: Supervised Incentive Spirometry (SIS)
- Non-Supervised Incentive Spirometry (Non-SIS) (Active Comparator): Participants perform incentive spirometry exercises independently using a provided guideline form. Supervisors provide daily reminders but do not directly observe the exercises. Participants log their activity daily.
  Interventions: Procedure: Non-Supervised Incentive Spirometry (Non-SIS)

INTERVENTIONS:
Procedure: Supervised Incentive Spirometry (SIS) — Participants perform incentive spirometry exercises twice daily for 3 days under direct supervision. The supervisor monitors technique, corrects errors, answers questions, and ensures exercises are done accurately. Each session includes 6 sets of 5 breaths, with slow inhalation, 2-second breath-hold, and slow exhalation, separated by rest periods. This intervention is performed in addition to standard cardiac rehabilitation.
  Arms: Supervised Incentive Spirometry (SIS)
Procedure: Non-Supervised Incentive Spirometry (Non-SIS) — Exercises independently using a guideline form with daily reminders. Participants log activity. 6 sets of 5 breaths per session.
  Arms: Non-Supervised Incentive Spirometry (Non-SIS)

SUMMARY:
This study aims to evaluate the effect of supervised incentive spirometry (SIS) compared to unsupervised incentive spirometry (Non-SIS) on pulmonary function in patients following coronary artery bypass graft (CABG) surgery. Participants perform incentive spirometry exercises twice daily for three days after extubation. Pulmonary function parameters, including forced expiratory volume in one second (FEV1), forced vital capacity (FVC), and peak expiratory flow (PEF), are assessed before and after the intervention period to compare changes between the two groups.

DETAILED DESCRIPTION:
Coronary artery bypass graft (CABG) surgery is associated with an increased risk of postoperative pulmonary complications, such as atelectasis, pneumonia, and pleural effusion, which may impair pulmonary function. Incentive spirometry (IS) is commonly used as part of postoperative care to promote deep breathing, enhance alveolar recruitment, and improve lung volumes.

This quasi-experimental study is conducted at Dr. Hasan Sadikin General Hospital, Bandung, Indonesia, and enrolls patients who have undergone CABG surgery. Participants are consecutively assigned to one of two intervention groups: supervised incentive spirometry (SIS) or unsupervised incentive spirometry (Non-SIS).

Participants in the SIS group perform incentive spirometry exercises under direct supervision by healthcare personnel twice daily to ensure correct technique and adherence. Participants in the Non-SIS group perform the same exercises independently with routine reminders. Both groups receive a standardized postoperative cardiac rehabilitation program.

Pulmonary function is assessed using a portable spirometer measuring forced expiratory volume in one second (FEV1), forced vital capacity (FVC), and peak expiratory flow (PEF). Measurements are conducted at 24 hours post-extubation (T1) and after three days of incentive spirometry exercises (T2). The primary objective is to compare changes in pulmonary function parameters between the supervised and unsupervised groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥18 years.
* Patients who have undergone Coronary Artery Bypass Graft (CABG) surgery.
* Mechanical ventilation <24 hours post-surgery.
* Physically able to perform incentive spirometry (IS) exercises.
* Signed informed consent to participate in the study.

Exclusion Criteria:

* Hemodynamically unstable patients.
* Patients with cognitive or communication impairments.
* Oral abnormalities that prevent the use of IS.
* Patients with Chronic Obstructive Pulmonary Disease (COPD).
* Patients with thoracic anomalies.
* Patients who required reintubation.
* History of incentive spirometry use within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 Second (FEV1) | T1 (24 hours post-extubation) and T2 (after 3 days of incentive spirometry exercise)
  Measures the volume of air that can be forcibly exhaled in one second to assess pulmonary function in post-CABG patients.

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) | T1 (24 hours post-extubation) and T2 (after 3 days of incentive spirometry exercise)
  Measures the total volume of air that can be exhaled after a maximal inhalation to evaluate restrictive ventilatory patterns in post-CABG patients.

OTHER OUTCOMES:
Peak Expiratory Flow (PEF) | T1 (24 hours post-extubation) and T2 (after 3 days of incentive spirometry exercise)
  Measures the maximal airflow during forced exhalation to assess the ability of the lungs to expel air in post-CABG patients.

CONTACTS AND LOCATIONS:
Locations (1):
- RSUP Dr. Hasan Sadikin, Bandung, West Java, Indonesia

REFERENCES:
- [Result] Ababneh QM, Abdelrahman H, Abdelhameed ME. Effectiveness of Incentive Spirometry Versus Deep Breathing Exercises in Preventing Postoperative Pulmonary Complications After Abdominal Surgery: A Comprehensive Review. Cureus. 2025 Mar 6;17(3):e80149. doi: 10.7759/cureus.80149. eCollection 2025 Mar. PMID 40190855
- [Result] do Nascimento Junior P, Modolo NS, Andrade S, Guimaraes MM, Braz LG, El Dib R. Incentive spirometry for prevention of postoperative pulmonary complications in upper abdominal surgery. Cochrane Database Syst Rev. 2014 Feb 8;2014(2):CD006058. doi: 10.1002/14651858.CD006058.pub3. PMID 24510642
- [Result] Alwekhyan SA, Alshraideh JA, Yousef KM, Hayajneh F. Nurse-guided incentive spirometry use and postoperative pulmonary complications among cardiac surgery patients: A randomized controlled trial. Int J Nurs Pract. 2022 Apr;28(2):e13023. doi: 10.1111/ijn.13023. Epub 2021 Oct 22. PMID 34676618
- [Result] Su H, Zhang J, Liu Y, Peng H, Zhang L. Pre and postoperative nurse-guided incentive spirometry versus physiotherapist-guided pre and postoperative breathing exercises in patients undergoing cardiac surgery: An evaluation of postoperative complications and length of hospital stay. Medicine (Baltimore). 2022 Dec 30;101(52):e32443. doi: 10.1097/MD.0000000000032443. PMID 36596066
- [Result] Melly L, Torregrossa G, Lee T, Jansens JL, Puskas JD. Fifty years of coronary artery bypass grafting. J Thorac Dis. 2018 Mar;10(3):1960-1967. doi: 10.21037/jtd.2018.02.43. PMID 29707352
- See also: Melly L, Torregrossa G, Lee T, Jansens JL, Puskas JD. Fifty years of coronary artery bypass grafting. J Thorac Dis. 2018;10(3):1960-7. — https://pubmed.ncbi.nlm.nih.gov/29707352/?utm_source=chatgpt.com
- See also: Su H, Zhang J, Liu Y, Peng H, Zhang L. Pre and postoperative nurse-guided incentive spirometry vs. physiotherapist-guided breathing exercises in cardiac surgery. Medicine (Baltimore). 2022;101(52):e32443. — https://pubmed.ncbi.nlm.nih.gov/36596066/?utm_source=chatgpt.com
- See also: Saja Ahmad Alwekhyan et al. Nurse-guided incentive spirometry use and postoperative pulmonary complications among cardiac surgery patients. Int J Nurs Pract. 2022;28(2):e13023. — https://pubmed.ncbi.nlm.nih.gov/34676618/?utm_source=chatgpt.com
- See also: do Nascimento Junior P, Módolo NS, Andrade S, Guimarães MM, Braz LG, El Dib R. Incentive spirometry for prevention of postoperative pulmonary complications in upper abdominal surgery. Cochrane Database Syst Rev. 2014;(2):CD006058.pub3. — https://pubmed.ncbi.nlm.nih.gov/24510642/?utm_source=chatgpt.com
- See also: Ababneh QM et al. Effectiveness of Incentive Spirometry Versus Deep Breathing Exercises in Preventing Postoperative Pulmonary Complications After Abdominal Surgery: A Comprehensive Review. Cureus. 2025;17(3):e80149. — https://pubmed.ncbi.nlm.nih.gov/40190855/?utm_source=chatgpt.com